CLINICAL TRIAL: NCT04644198
Title: Pilot Study of Convalescent COVID-19 Plasma Transfusion in Severe COVID-19 Patients at a Type A Teaching Hospital in Jamaica
Brief Title: Convalescent Plasma Transfusion in Severe COVID-19 Patients in Jamaica
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of The West Indies (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ECP/195,19/20
Record Dates: First submitted 2020-11-18; First posted 2020-11-25 (Actual); Last update posted 2021-05-12 (Actual); Status verified 2020-11

CONDITIONS: COVID-19, Convalescent Plasma Treatment
Keywords: Donor; Recipients; Transfusion; Convalescent plasma; COVID Viral Load
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Convalescent Plasma Treatment (Active Comparator): Convalescent Plasma
  Interventions: Biological: Convalescent Plasma Infusion
- Control (No Intervention): Standard of care

INTERVENTIONS:
Biological: Convalescent Plasma Infusion — 250 mls of convalescent plasma on day 1 & 2.
  Arms: Convalescent Plasma Treatment

SUMMARY:
Corona virus Disease 2019 (COVID-19) can be a severe respiratory illness caused by Severe Acute Respiratory Syndrome (SARS-CoV2) for which there is no standard treatment in affected persons nor a vaccine to prevent the infection. The investigators propose to test whether the use of Convalescent plasma given to patients with severe COVID-19 disease will decrease risk of death, decrease use of ventilatory support decrease biomarkers of inflammation and improve measures of viral replication compared with controls subjects who were not transfused.Convalescent plasma, will be collected from persons who are more than 21 days post negative viral testing or 28 days post resolution of symptoms.

DETAILED DESCRIPTION:
Coronavirus Disease 2019 (COVID-19) can be a severe respiratory illness caused by SARS-CoV2 for which there is no standard treatment in affected persons nor a vaccine to prevent the infection. This condition has and continues to cause significant burden on Health care systems with affected persons needing prolonged stay on ventilators in Intensive Care Units.

Convalescent plasma has been used in the treatment of other life-threatening conditions such as Novel Influenza A (H1N1) pandemic, SARS-COV-1 epidemic and Middle East respiratory syndrome -related Coronavirus (MERS-CoV) epidemic. Since convalescent plasma has been found to be beneficial in some diseases but is not always successful in all conditions in which it has been tried, there is no guarantee of success in this disease, and so it is necessary to conduct this study.

A sample of 30 patients with severe and life threatening COVID-19 disease will participate in phase 2 clinical trials. Convalescent Plasma will be administered to participants fulfilling the criteria due to its proven effect on H1N1 pandemic, SARS-COV-1 and MERS-COV epidemic. Although it has proven beneficial in some diseases, there is no guarantee that it will bring the desired outcome , hence the importance of the clinical trials. The observation will consist of three groups, namely, donor, participants and a control group. These patients must recover from all COVID-19 symptoms.

The participants who fulfill the inclusion criteria will receive convalescent plasma, collected from persons who are more than 21 days post negative viral testing or 28 days post resolution of symptoms. Potential participants will be approached by a research assistant within 24 hours of diagnosis and be told about the study and informed consent obtained only after the participants are identified as meeting the inclusion criteria for either participation as donor or recipient of plasma. If in the case of recipients, the recipients are intubated or otherwise unable to give consent, the recipients proxy will be required to do the same before participation is allowed. Plasma donations will also be solicited on the University of the West Indies (UWI) and University Hospital of the West Indies (UHWI) websites and Mona Messaging platform of UWI as well as social media platforms that will be managed by the UHWI public relations department. In addition, the investigators will also use electronic news media publications to inform interested persons about the study.

A sample of the recipients plasma will be kept for future studies as yet unknown. If any of these are genetic studies, attempts will be made to re-contact the donors to consent to these studies. The duration for this first study will be for one year.

The recipients for this plasma infusion must fulfill criteria for severe or immediately life-threatening infection. The control group will also fulfill the criteria for severe or life-threatening disease but have a contraindication to receiving plasma. The plasma donors must fulfill the criteria for selection of blood donors but in addition would have been recovered from COVID-19.

The data analysis will include changes in means of the objectives using Student's t-test.

Each participant will be assigned a study identification (ID) number and data linked to the study ID will only be accessible to researchers using a password protected computer.

The participants name and study ID number will be kept in a locked filing cabinet with access only to the research team.

This is a moderate risk study and participants will be informed that no personal benefit will be derive from participating in this study.

Limitations include not getting enough persons for plasma donation if the infection rate in Jamaica remains low, or the age of the affected persons is outside of the accepted range of our blood donor requirements. As this is a pilot however, the investigators may be able to achieve the sample size which should allow the investigators to identify any challenges in conducting a larger trial.

Participants will have every effort made to maintain confidentiality by using only study ID numbers on data collection sheets and laboratory studies.

ELIGIBILITY:
Inclusion Criteria

* 18 years of age or older:
* Laboratory confirmed COVID-19:
* Severe or immediately life-threatening COVID-19:
* Severe disease is defined as one or more of the following:

Exclusion Criteria:

* Patients with mild or moderate COVID-19 infection that do not need in-patient care:
* Patients with a history of severe allergic reaction to plasma infusion:
* Patients who do not give consent or withdraw consent from study:

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2021-12-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Mortality | Time from Admission up 28 days post-discharge
  Number of deaths
Viral load | Change in viral titres up to 28 days after transfusion measured on day 1, 3, 5, 7, 14, 28 after receiving transfusion
  COVID-19 Viral titres
Antibody titre for Immunoglobulin (IgG) anti-SARS-CoV-2 antibody | Change in antibody titres up to 28 days after transfusion measured on day 1, 3, 5, 7, 14, 28 after receiving transfusion
  Antibody titre for IgG anti-SARS-CoV-2 antibody
Antibody titre for Immunoglobulin A (IgA) anti-SARS-CoV-2 antibody | Change in antibody titres up to 28 days after transfusion measured on day 1, 3, 5, 7, 14, 28 after receiving transfusion
  Antibody titre for IgA anti-SARS-CoV-2 antibody
Procalcitonin titres | Change in titres up to 28 days after transfusion measured on day 1, 3, 5, 7, 14, 28 after receiving transfusion
  Procalcitonin levels
Interleukin 6 (IL-6) | Change in titres up to 28 days after transfusion measured on day 1, 3, 5, 7, 14, 28 after receiving transfusion
  Interleukin 6 (IL-6) levels
D-dimer | Change in titres up to 28 days after transfusion measured on day 1, 3, 5, 7, 14, 28 after receiving transfusion
  D-dimer levels
C-reactive protein | Change in titres up to 28 days after transfusion measured on day 1, 3, 5, 7, 14, 28 after receiving transfusion
  C- reactive protein levels
Ferritin | Change in titres up to 28 days after transfusion measured on day 1, 3, 5, 7, 14, 28 after receiving transfusion
  Ferritin levels

SECONDARY OUTCOMES:
Length of ICU admission | Number of days from hospital admission up to day of discharge assessed up to 100 days
  Duration of stay in ICU
Days to recovery | Number of days from hospital admission up to the day of recovery assessed up to 100 days
  Time to recovery

CONTACTS AND LOCATIONS:
Overall Officials: Gilian G Wharfe, Principal Investigator — University of the West Indies
Locations (1):
- University of the West Indies, Kingston, Jamaica